CLINICAL TRIAL: NCT03878004
Title: A Double-blind, Randomized, Multicentre, Placebo-controlled Phase II Clinical Trial of Safety and Immunogenicity of Recombinant Subunit Tuberculosis Vaccine GamTBvac in Healthy Adults
Brief Title: Phase II Clinical Trial of Safety and Immunogenicity of Recombinant Subunit Tuberculosis Vaccine GamTBvac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: contract research organization Cromos Pharma (Unknown); contract research organization K-Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-GamTBvac-2018
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Tuberculosis; Mycobacterium tuberculosis; Recombinant vaccine; Mycobacterium Infections; Vaccines
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized (in 3:1 ratio -vaccine : placebo) study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Group (Experimental): 135 people who will receive the vaccine in the therapeutic scheme
  Interventions: Biological: GamTBvac vaccine
- Placebo Group (Placebo Comparator): 45 people who will receive placebo in the therapeutic scheme
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: GamTBvac vaccine — introduction of GamTBvac (lyophilisate for preparation of solution for subcutaneous administration, 5.35 mg / dose) twice into a shoulder with an 8-week interval.
  Arms: Primary Group
Biological: placebo — introduction of placebo twice into a shoulder with an 8-week interval.
  Arms: Placebo Group

SUMMARY:
This is a double-blind, randomized (in 3:1 ratio -vaccine : placebo) study to assess the safety, reactogenicity and immunogenicity in healthy, BCG vaccinated adults.

DETAILED DESCRIPTION:
Participants will be randomized in two groups (in 3:1 ratio -vaccine : placebo) to receive two doses of either GamTBvac or placebo. Subjects will be followed for 5 months after dose 1.

The primary goal of this study is to assess the immunogenicity of a tuberculosis subunit recombinant GamTBvac vaccine in a vaccination scheme with double administration to healthy volunteers.

The secondary goal of this study is the in-depth assessment of the safety and reactogenicity of the tuberculosis subunit recombinant vaccine GamTBvac when given twice to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study requirements, sign the Informed Consent Form (ICF) and consent to all restrictions applicable during the study.
2. Participants must be 18 to 49 years of age inclusive, at the time of signing the informed consent.
3. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination and laboratory tests.
4. No evidence of pulmonary pathology as confirmed by chest X-ray.
5. Body Mass Index (BMI) 18 to 30 kg/m2, inclusive.
6. Male and female.
7. For female participants: a female participant is eligible to participate if she is not pregnant (has a negative pregnancy test (dipstrip) at screening and at Study Day 0), not breastfeeding, and at least one of the following conditions applies: a) Not a women of childbearing potential (WOCBP) OR b) A WOCBP who agrees to follow the contraceptive guidance during the full duration of the study.
8. Had BCG vaccination, documented through medical history or presence of scar.
9. Positive result of PPD-L test: induration 5 mm and 9 mm.
10. The absence of markers of the immune response to mycobacterial proteins ESAT6 and CFP10, which characterize the probable contact with M. tuberculosis preceding the beginning of the study in Diaskintest and QuantiFERON TB Gold ELISA tests at the same time on screening.
11. The absence of the fact of living or working with someone who has a diagnosis of tuberculosis for 3 months before Day 0 of the study.
12. The absence of malignant neoplasms at the moment and for 5 years before being included in the study.
13. The absence of malignant blood diseases.

Exclusion Criteria:

1. The presence of symptoms of acute illness, including the temperature in the axillary cavity of more than 37.5 C, for 5 days before the start of the study and on day 0 of the study.
2. Anamnesis or the presence of tuberculosis, including extrapulmonary tuberculosis.
3. Negative result of PPD-L test ( less than 5 mm) or hyperergic positive PPD-L test (more than 9 mm).
4. The presence of a positive or doubtful result in the tests Diaskintest and / or QuantiFERON TB Gold ELISA.
5. Anamnesis or the presence of autoimmune diseases or immunosuppression, or a family history of congenital or hereditary immunodeficiency.
6. Positive tests for the presence of HIV-1/2 antibodies, HBsAg or hepatitis C antibodies on screening.
7. Use of immunosuppressive or other immunomodulatory drugs for 42 days before Day 0 of the study.
8. Use of immunoglobulin or blood products for 180 days prior to Day 0 of the study or a plan for their appointment during the study.
9. Use of any study drug or vaccine under study for 90 days prior to the day of screening, or planned participation in other clinical studies during the study.
10. Use of antibacterial drugs within 14 days prior to Day 0 of the study (oral administration) or within 28 days before Day 0 of the study (parenteral administration).
11. Use the tested GamTBvac at any time before day 0 of the study.
12. Planned use / prescription of a registered vaccine within 28 days before and 28 days after vaccination with the vaccine in question.
13. Planned surgery (in a planned manner) during the study.
14. Anamnesis or presence according to laboratory data of any possible immunodeficiency state.
15. A history of allergic diseases or reactions that may be aggravated by any component of the vaccine in question.
16. The medical history of diseases that may endanger the safety of the participant, including but not limited to: deterioration of lung function in any lung disease, heart or kidney failure, neurological diseases, epilepsy or infant convulsions, diabetes, cancer.
17. Anamnesis or the presence of any systemic diseases or any chronic diseases that, in the opinion of the researcher, may affect the safety assessment or the reactogenicity or immunogenicity of the vaccine under investigation.
18. Anamnesis of chronic abuse of alcohol or drugs.
19. Anamnesis or the presence of diseases or features of the skin, which, according to the researcher, may affect the evaluation of reactions at the injection site (diseases: malignant skin, allergic and eczematous skin diseases; features: congenital or acquired benign lesions on the skin (nevus) , scars, decorative modifications of the body (applying a permanent (resistant) pattern, tattoos) applied drawings).
20. Volunteer participation in any other clinical study over the past 90 days.
21. Donor blood donation (450 ml or more of blood or plasma) less than 2 months prior to inclusion in the study.
22. The presence of allergic reactions to animal proteins and a tuberculin allergen in history.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
level of IFN-y secretion in whole blood or PBMC fraction | Day 0 through month 5
  1. Secretion level of IFN-y by whole blood or PBMC fraction in response to stimulation with vaccine antigens
Number of Participants With Adverse Events | Day 1 - month 5
  Determining the frequency of an undesirable immediate response response within 2 hours after vaccine administration; assessment of the frequency of local and systemic requests for the entire observation period after the 1-st vaccination and the 2-nd vaccination

SECONDARY OUTCOMES:
CD4+ and CD8+ T cells | Day 0 through month 5
  Percentage of CD4+ and CD8+ T cells that express IFN-y, TNF, and/or IL-2 alone or in combination in response to stimulation with vaccine antigens (representing the full sequence of the vaccine antigens or its separate domains)
titer of antibodies of the IgG class | Day 0 - month 5
  A change in the titer of antibodies of the IgG class (induction of the humoral response) to the complete sequence of vaccine antigens or their individual domains, determined using multiplex suspension enzyme immunoassay timeline.
QuantiFERON TB | Day 0, month 5
  A positive result in the quantum test using the QuantiFERON TB Gold ELISA reagent kit.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - "City polyclinic № 2 Of the Department of health of the city of Moscow", Выделите текст, чтобы посмотреть примеры, Moscow
  - Sechenov University, Moscow

IPD SHARING:
Plan to Share IPD: Undecided